CLINICAL TRIAL: NCT06535334
Title: Intravenous Chemotherapy Versus Intraperitoneal Chemotherapy in Recurrent Ovarian Cancer
Brief Title: Intraperitoneal Chemotherapy in Recurrent Ovarian Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Professor, Far Eastern Memorial Hospital
Other Study IDs: 113130-E
Record Dates: First submitted 2024-06-06; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Intravenous Chemotherapy Versus Intraperitoneal Chemotherapy in Recurrent Ovarian Cancer
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intravenous chemotherapy: triweekly chemotherapy with carboplatin AUC=5~6 + liposomal-doxorubicin 30~40mg/m2 or paclitaxel 175mg/m2 0r docetaxel 60~75mg/m2
  Interventions: Drug: Chemotherapy
- intraperitoneal chemotherapy: Day 1 IV Paclitaxel 135 mg/m2 + IP Cisplatin 75-100 mg/m2 or IP carboplatin (AUC = 6) Day 8 IP Paclitaxel 60 mg/m2 Every 21 days * 6 cycles
  OR
  Day 1 IP Carboplatin AUC=5 or IP Cisplatin 50-75mg/m2 Day 2 IV Liposomal doxorubicin 15 mg/m2 + IP Liposomal doxorubicin 15 mg/m2 Every 28 days * 6 cycles
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Intravenous chemotherapy versus intraperitoneal chemotherapy in recurrent ovarian cancer

SUMMARY:
This study aims to compare intravenous chemotherapy versus intraperitoneal chemotherapy in patients with recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* women who had recurrent ovarian cancer and was treated with either intravenous or intraperitoneal platinum based chemotherapy

Exclusion Criteria:

* women who did not complete the designated treatment course (exception to those who had to quit due to progressive disease or death of any cause)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with ovarian cancer
Study Population: woman with recurrent ovarian cancer who was treated with chemotherapy (either intravenous or intraperitoneal)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
RFS | the time interval from the date of surgery or the start of chemotherapy to clinically defined recurrence, disease progression, death from any cause or last follow-up
  Recurrence free survival
OS | the time interval from the date of surgery or the start of chemotherapy to the date of death from any cause or last follow-up
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No